CLINICAL TRIAL: NCT01777503
Title: Phase IV: A Comparison of Reduced-dose Prasugrel and Clopidogrel in Elderly Patients With Acute Coronary Syndrome Undergoing Early Percutaneous Coronary Intervention (PCI)
Brief Title: The Elderly ACS II Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: ANMCO Italian Association of Hospital Cardiologist (Unknown); Italian Society of Invasive Cardiology (Other); A. Manzoni Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT Number: 2012-002882-37
Record Dates: First submitted 2013-01-21; First posted 2013-01-29 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome; Coronary Arteriosclerosis; Myocardial Ischemia; Cardiovascular Diseases
Keywords: acute coronary syndrome; elderly; percutaneous revascularization; antiaggregant drugs
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prasugrel (Experimental): prasugrel 60 mg loading dose, followed by 5 mg once daily until the end of follow-up
  Interventions: Drug: prasugrel
- clopidogrel (Active Comparator): Clopidogrel 300 mg loading dose followed by 75 mg once day until the end of follow-up
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: prasugrel — prasugrel 5 mg o.d.
  Other Names: Efient
  Arms: prasugrel
Drug: Clopidogrel — 75 mg o.d.
  Other Names: Plavix
  Arms: clopidogrel

SUMMARY:
The objective of this study is to compare reduced-dose prasugrel and standard dose clopidogrel in patients older than 74 years with ACS, including non-ST-elevation (NSTEACS) and ST-elevation (STEMI) patients, undergoing early PCI. The primary endpoint of the trial will be the one-year composite of (all-cause)death, myocardial infarction, stroke and re-hospitalization due to cardiovascular reasons or bleeding.

ELIGIBILITY:
Inclusion Criteria:

- Patients >74 years of age hospitalized for an ACS, with or without STE, with an onset of symptoms during the previous 72 hours, and candidates to an early PCI.

* STEMI patients may be randomized upon first diagnosis, provided they do not meet any exclusion criteria. STEMI patients should not exceed 50 percent of the global population of the study
* Eligible NSTEACS patients may be randomized after coronary angiography. To be eligible, NSTEACS patients must have at least one of the following characteristics:

  * elevated troponin levels;
  * diabetes mellitus;
  * prior MI;
  * at least one new ischemic episode while on standard treatment during the index hospitalization;
  * ACS due to stent thrombosis.

Exclusion Criteria:

* History of stroke or transient ischemic attack (TIA)
* Gastrointestinal or genitourinary bleeding of clinical significance within 6 weeks prior to randomization.
* Hemoglobin level on admission <10 g/dl, unless this is considered to be secondary to renal dysfunction or known myelodysplasia.
* Secondary causes of acute myocardial ischemia.
* Known current platelet count < 90,000 cells/mL.
* Ongoing oral anticoagulant treatment or an INR known to be >1.5 at the time of screening.
* Concomitant severe obstructive lung disease, malignancy or neurologic deficit limiting follow-up or adherence to the study protocol.
* Participation in any phase of another clinical research study involving the evaluation of another investigational drug or device within 30 days prior to randomization
* Inability to give at least verbal informed consent to the study.
* Contraindications to the use of clopidogrel or prasugrel as per package leaflet.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1457 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
The composite of all-cause mortality, myocardial infarction (MI), disabling stroke and re-hospitalization for cardiovascular causes or bleeding within one year | 1 year

SECONDARY OUTCOMES:
The composite of burden of recurrent cardiovascular (CV) events, CV mortality, all-cause mortality and MI, major bleeding, any stroke, total number of days spent in hospital. | 1 year
  definition of major bleeding:
  - Bleeding Academic Research Consortium (BARC) type 2 or 3 bleeding within 1 year (for bleedings occurring during index or subsequent hospitalizations)
  · BARC type IV bleeding within 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Arcispedale Santa Maria Nuova- IRCCS, Reggio Emilia, Italy
  - Azienda Ospedaliera "Ospedale Civile di Legnano", Legnano, MI

REFERENCES:
- [Derived] Crimi G, Morici N, Ferrario M, Ferri LA, Piatti L, Grosseto D, Cacucci M, Mandurino Mirizzi A, Toso A, Piscione F, De Carlo M, Elia LR, Trimarco B, Bolognese L, Bovenzi FM, De Luca G, Savonitto S, De Servi S. Time Course of Ischemic and Bleeding Burden in Elderly Patients With Acute Coronary Syndromes Randomized to Low-Dose Prasugrel or Clopidogrel. J Am Heart Assoc. 2019 Jan 22;8(2):e010956. doi: 10.1161/JAHA.118.010956. PMID 30636561
- [Derived] Savonitto S, Ferri LA, Piatti L, Grosseto D, Piovaccari G, Morici N, Bossi I, Sganzerla P, Tortorella G, Cacucci M, Ferrario M, Murena E, Sibilio G, Tondi S, Toso A, Bongioanni S, Ravera A, Corrada E, Mariani M, Di Ascenzo L, Petronio AS, Cavallini C, Vitrella G, Rogacka R, Antonicelli R, Cesana BM, De Luca L, Ottani F, De Luca G, Piscione F, Moffa N, De Servi S; Elderly ACS 2 Investigators. Comparison of Reduced-Dose Prasugrel and Standard-Dose Clopidogrel in Elderly Patients With Acute Coronary Syndromes Undergoing Early Percutaneous Revascularization. Circulation. 2018 Jun 5;137(23):2435-2445. doi: 10.1161/CIRCULATIONAHA.117.032180. Epub 2018 Feb 19. PMID 29459361
- [Derived] Ferri LA, Morici N, Grosseto D, Tortorella G, Bossi I, Sganzerla P, Cacucci M, Sibilio G, Tondi S, Toso A, Ferrario M, Gandolfo N, Ravera A, Mariani M, Corrada E, Di Ascenzo L, Petronio AS, Cavallini C, Moffa N, De Servi S, Savonitto S. A comparison of reduced-dose prasugrel and standard-dose clopidogrel in elderly patients with acute coronary syndromes undergoing early percutaneous revascularization: Design and rationale of the randomized Elderly-ACS 2 study. Am Heart J. 2016 Nov;181:101-106. doi: 10.1016/j.ahj.2016.08.010. Epub 2016 Aug 26. PMID 27823681
- See also: Design and rationale of the randomized Elderly-ACS 2 study — http://dx.doi.org/10.1016/j.ahj.2016.08.010